CLINICAL TRIAL: NCT01634750
Title: A Phase 1 Randomized, Placebo-Controlled, Double-Blind, Escalating Single-Dose Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of ManNAc in Subjects With GNE Myopathy or Hereditary Inclusion Body Myopathy (HIBM)
Brief Title: Phase I Clinical Trial of ManNAc in Patients With GNE Myopathy or Hereditary Inclusion Body Myopathy (HIBM)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH); Therapeutics for Rare and Neglected Diseases (TRND) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 120207; 12-HG-0207
Record Dates: First submitted 2012-07-03; First posted 2012-07-06 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-02-24

CONDITIONS: Hereditary Inclusion Body Myopathy (HIBM); GNE Myopathy
Keywords: N-Acetyl-D-mannosamine (ManNAc); HIBM; GNE Myopathy
MeSH Terms: conditions — Distal myopathy, Nonaka type | interventions — N-acetylmannosamine

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- ManNac (Experimental)
  Interventions: Drug: ManNAc
- Placebo (Placebo Comparator)
  Interventions: Drug: ManNAc

INTERVENTIONS:
Drug: ManNAc — Single dose

SUMMARY:
Background:

- Hereditary inclusion body myopathy (HIBM) is a genetic disorder caused by mutations in a gene called GNE. This gene is responsible for producing a sugar called sialic acid. Low levels of sialic acid may cause muscle problems. Symptoms of HIBM include walking difficulties and muscle weakness, which usually start in a person s 20s or 30s and become worse over time.

Researchers are studying a drug called ManNAc. It may be useful for treating HIBM. However, this drug is still being tested. Researchers want to see how ManNAc is absorbed into and removed from the blood. They will not be looking specifically at whether ManNAc can stop or slow the symptoms of HIBM.

Objectives:

* <TAB>To study how MaNAc is absorbed into and removed from the blood in people with HIBM.
* <TAB>To study of safety of ManNAc in people with HIBM.

Eligibility:

- Individuals between 18 and 70 years of age who have HIBM.

Design:

* Participants will be screened with a physical exam and medical history. Blood and urine samples will be collected.
* Participants will have a 3 to 4-day inpatient stay for the main part of the study.
* Participants will be divided into groups of six. In each group, four will take ManNAc and two will take a placebo. Participants will not know which one they will receive.
* Participants will have a single dose of either ManNAc or placebo. They will be monitored for any possible side effects. Frequent blood samples will be collected during the 4-day stay.
* No treatment for HIBM will be provided as part of this study.

DETAILED DESCRIPTION:
Hereditary inclusion body myopathy (HIBM) is an autosomal recessive, neuromuscular disorder characterized by progressive muscle weakness with onset in early adulthood. The causative gene, GNE, codes for the bifunctional enzyme uridine diphospho-N-acetylglucosamine (UDP-GlcNAc)-2-epimerase/N-acetylmannosamine (ManNAc) kinase (GNE/MNK), which catalyzes the first 2 steps in the biosynthesis of sialic acid. The subsequent paucity of sialic acid production is presumed to cause decreased sialylation of HIBM muscle glycoproteins, resulting in muscle deterioration. In this Phase 1, randomized, placebo-controlled, double-blind, escalating single-dose study, we propose to provide ManNAc (N-acetyl-D-mannosamine monohydrate) orally as a liquid solution to 3 cohorts of 6 subjects (Cohorts A, B, C) at doses of 3,000 mg, 6,000 mg, and 10,000 mg ManNAc, respectively, or up to the maximum tolerated dose (MTD). The objectives of this study are to evaluate the safety, tolerability, and pharmacokinetics (PK) of a single dose of orally administered ManNAc to HIBM subjects, to identify the MTD of a single dose of orally administered ManNAc to HIBM subjects, and to explore the effect of a single dose of ManNAc on potential pharmacodynamic (PD) markers of HIBM. All subjects will be randomly assigned in a 2:1 ratio to receive ManNAc (n equals 4) or placebo (n equals 2) and the decision to dose-escalate will be the responsibility of the Safety Review Committee (SRC). Safety will be assessed by adverse events (AEs), clinical laboratory tests, vital signs, physical examinations, and electrocardiograms (ECGs). PK will be assessed for both ManNAc and sialic acid.

ELIGIBILITY:
* INCLUSIONI CRITERIA:
* Subject is 18-70 years, either gender, inclusive.
* Subject has a diagnosis of HIBM (or IBM2, GNE myopathy, DMRV or Nonaka myopathy) based upon a consistent clinical course and identification of 2 GNE mutations. Molecular confirmation of the diagnosis will be obtained for all subjects in the study.
* Subject must be willing to stop any treatment with ManNAc, sialic acid, IVIG, and/or other supplements containing sialic acid (eg, St John s wort, sialyllactose) 30 days prior to randomization and remain off such treatment for the duration of the trial.
* Subject has the ability to travel to the NIH Clinical Center (CC) for admissions.
* Subject (if a woman of reproductive age) must be willing to use an effective method of contraception for the duration of the trial.
* Subject provides written informed consent.

EXCLUSION CRITERIA:

* Subject has a severe disease manifestation that would interfere with the ability to comply with the requirements of this protocol.
* Subject has a psychiatric illness or neurological disease that would interfere with the ability to comply with the requirements of this protocol. This includes, but is not limited to, uncontrolled/untreated psychotic depression, bipolar disorder, schizophrenia, substance abuse or dependence, antisocial personality disorder, or panic disorder.
* Subject has hepatic laboratory parameters (AST, ALT, GGTP), or renal laboratory parameters (creatinine, BUN) greater than 3 times the upper limit of normal.
* Subject has a QTcB >450 msec (males) or QTcB >470 msec (females).
* Subject is anemic (defined as two standard deviations below normal for age and gender).
* Subject shows evidence of clinically significant cardiovascular, pulmonary, hepatic, renal, hematological, metabolic, or gastrointestinal disease, or has a condition that requires immediate surgical intervention.
* Subject is pregnant or breastfeeding at any time during the study.
* Subject has received treatment with another investigational drug, investigational device, or approved therapy for investigational use within 4 weeks of initial screening.
* Subject has a hypersensitivity to ManNAc or in the judgment of the investigator, has a condition that places the subject at increased risk for adverse effects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09-11; Study Completion 2013-05-29 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of a single dose of orally administered ManNAc to HIBM subjects.

SECONDARY OUTCOMES:
Pharmacokinetics

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Carrillo-Carrasco, M.D., Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Amir SM, Barker SA, Butt WR, Crooke AC, Davies AG. Administration of N-acetyl-D-mannosamine to mammals. Nature. 1966 Aug 27;211(5052):976-7. doi: 10.1038/211976a0. No abstract available. PMID 5970419
- [Background] Argov Z, Mitrani-Rosenbaum S. The hereditary inclusion body myopathy enigma and its future therapy. Neurotherapeutics. 2008 Oct;5(4):633-7. doi: 10.1016/j.nurt.2008.07.004. PMID 19019317
- [Background] Bork K, Reutter W, Gerardy-Schahn R, Horstkorte R. The intracellular concentration of sialic acid regulates the polysialylation of the neural cell adhesion molecule. FEBS Lett. 2005 Sep 12;579(22):5079-83. doi: 10.1016/j.febslet.2005.08.013. PMID 16137682
- [Derived] Van Wart S, Mager DE, Bednasz CJ, Huizing M, Carrillo N. Population Pharmacokinetic Model of N-acetylmannosamine (ManNAc) and N-acetylneuraminic acid (Neu5Ac) in Subjects with GNE Myopathy. Drugs R D. 2021 Jun;21(2):189-202. doi: 10.1007/s40268-021-00343-6. Epub 2021 Apr 24. PMID 33893973
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-HG-0207.html